CLINICAL TRIAL: NCT04468698
Title: Intra-Abdominal Pressure Effect on Intra-Abdominal Volume and Airway Pressures During Pneumoperitoneum Insufflation - a Patient-Level Meta-Analysis of Three Randomized Clinical Trials
Brief Title: Intra-Abdominal Pressure Effect on Intra-Abdominal Volume and Airway Pressures During Laparoscopy
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator, Hospital Universitario La Fe
Other Study IDs: VoIPP
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Surgery; Pneumoperitoneum; Intra Abdominal Pressure
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Global cohort: A global cohort is built merging data from three studies
  Interventions: Other: Peritoneum insufflation

INTERVENTIONS:
Other: Peritoneum insufflation — Before surgery pneumoperitoneum is established by insufflating gas into the abdomen. Intraabdominal pressure (IAP) is set to 15 mmHg for initial abdominal stretching and then decreased in a stepwise manner down until 8 mmHg.

SUMMARY:
During pneumoperitoneum insufflation the insufflated gas increase intra-abdominal pressure. The generated pressure can lead to a different increase in volume depending on the abdominal cavity and patients' characteristics.

The primary objective is to determine the relationship between intraabdominal pressure (IAP) and intraabdominal volume (IAV) during pneumoperitoneum insufflation. The secondary objective is to determine the rate of abdominal-thoracic transmission (ATT) assessing the correlation between IAP and respiratory driving pressure (ΔPRS).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled one of the three studies (IPPCollapse I, II or III).
* underwent an initial insufflation procedure with a stepwise change in intraabdominal pressure to record Intraabdominal volume
* data from insufflation at 5 cmH2O of PEEP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing pneumoperitoenum insufflation during general anesthesia and mechanical venitlation.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Intraabdominal volume | During pneumoperitoneum insufflation before surgery

SECONDARY OUTCOMES:
Driving pressure | During pneumoperitoneum insufflation before surgery
  This is the pressure that exert a stress on the respiratory system during mechanical ventilation. It is calculated by subtracting the positive endexpiratory pressure from plateau pressure
Plateau pressure | During pneumoperitoneum insufflation before surgery
  This is the pressure in the airway during the mechanical venitilation inspiratory pause time

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital la Fe, Valencia, Spain